CLINICAL TRIAL: NCT05130697
Title: A Multicenter Survey Study Into Patient Experience With Mobile Apps
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University of Ireland, Galway, Ireland (Other)
Responsible Party: Principal Investigator, Michelle Tierney, Principal Investigator, National University of Ireland, Galway, Ireland
Other Study IDs: 2020.10.024; 2020-1089 (Other: The University of Texas MD Anderson Cancer Center)
Record Dates: First submitted 2021-11-05; First posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Malignant Pleural Effusion
MeSH Terms: conditions — Pleural Effusion, Malignant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: eMPowEr App — A mobile app to support participants in the management of malignant pleural effusions at home

SUMMARY:
This multicenter prospective survey study is designed to evaluate a newly developed mobile app that will support patients with malignant pleural effusion (MPE) treated with an indwelling pleural catheter (IPC). The aim is to test the mobile app with patients with MPE and get user feedback during and at the end of the study period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with MPE and, scheduled for an indwelling pleural catheter (IPC) procedure,
* Age 18 or older

Exclusion Criteria:

* Patients without an iOS smartphone or email account
* Patients who refuse participation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants (patients with MPE and an IPC in place) are being requested to use a pilot mobile app that is being developed to support them in their symptom management at home and to provide feedback on its usability.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
The % positive usability rating rated via an mHealth App Usability Questionnaire (MAUQ) | 2 weeks
  The % positive usability rating rated via an mHealth App Usability Questionnaire (MAUQ)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Galway, Galway, Ireland